CLINICAL TRIAL: NCT03644225
Title: Mechanical Characterization of Healthy and Diseased Skin With Suction Based Assessment of Skin Deformability
Brief Title: Suction Based Characterization of Healthy and Diseased Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oliver Distler (Other)
Collaborators: Swiss Federal Institute of Technology (Other)
Responsible Party: Sponsor-Investigator, Oliver Distler, Prof.Dr.med.Oliver Distler, Director of the Department of Rhumatology, University Hospital Zurich, University of Zurich
Organization: University of Zurich (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Swissmedic:2017-MD_0045; 2017-01154 (Other: Ethikkommission)
Record Dates: First submitted 2018-05-04; First posted 2018-08-23 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Intervention Model Description: Primary outcome:
  Mechanical characterization of healthy and diseased skin using novel aspiration device and comparing it to the already validated Cutometer® MPA 580. Comparison of mechanical skin properties of healthy to patients' skin tissue (control vs. examined group).
  Secondary outcome:
  Defining predictors of the skin worsening.
Masking Description: No randomisation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Control (Other): Healthy controls, who signed an informed consent, age ≥18 years old will be age and sex matched to the SSc patients
  Interventions: Device: Measurment with Aspirational Medical Device; Device: Measurment with Cutometer MPA 580
- Systemic sclerosis patients (Other): SSc patients who signed an Informed consent
  * Age ≥18 years old
  * Diagnosis of systemic sclerosis according to the ACR/EULAR 2013 criteria
  * Skin thickening diagnosed by clinical expert
  Interventions: Device: Measurment with Aspirational Medical Device; Device: Measurment with Cutometer MPA 580

INTERVENTIONS:
Device: Measurment with Aspirational Medical Device — The mechanical properties of healthy and SSc-diseased skin will be assessed by suction based measurements with a new developed Aspirational Medical Device.
Device: Measurment with Cutometer MPA 580 — The mechanical properties of healthy and SSc-diseased skin will be assessed by CE-marked Cutometer MPA 580

SUMMARY:
The mechanical properties of healthy and SSc-diseased skin will be assessed by suction based measurements. The negative pressure needed to gain a certain tissue elevation, tissue elevation in response to a certain negative pressure as well as the time of retraction of tissue will be recorded and analyzed. Mesurments will be done with the new developed Aspiration Device_Nimble and with the CE-certified Cutometer MPA 580.

DETAILED DESCRIPTION:
Patients with systemic sclerosis (SSc) show a thickening of the skin due to massive deposition of collagen and temporary edema in the dermis. The clinical palpation method is currently the only diagnosis method. For an objective detection a non-invasive skin elasticity measurement can be performed. The widely used approach is based on local tissue suction. This study aims at an identification and quantification of mechanical and structural properties of human skin. The results will then be compared in age- and gender matched control groups. For evaluation of the skin elasticity measurement the results will be compared to the clinical parametar validated, modified Rodnan skin score (mRSS).

The mechanical properties of healthy and diseased skin will be assessed by suction based measurements. The negative pressure is needed to gain a certain tissue elevation. Tissue elevation in response to a certain negative pressure as well as the time of retraction of tissue will be recorded and analyzed. (The different parameters depend on

ELIGIBILITY:
Inclusion Criteria:

-Signed Informed Consent

Healthy volunteers:

- Age ≥18 years old

SSc-Patients:

* Age ≥18 years old
* Diagnosis of systemic sclerosis according to the ACR/EULAR 2013 criteria
* Skin thickening diagnosed by clinical expert

Exclusion Criteria:

* Known or suspected non-compliance, drug or alcohol abuse,
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Previous enrolment into the current study,
* Participants, who are unable to hold still
* Impaired skin at the regions of measurements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 67 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2019-06-04 (Actual); Study Completion 2019-06-04 (Actual)

PRIMARY OUTCOMES:
Mechanical characterization of healthy and diseased skin using novel aspiration device and comparing it to the already validated Cutometer® MPA 580. | one visit, one measurement, one year
  The stiffness (mbar/mm) properties of healthy skin and SSc skin will be measured with the Aspiration Device and the Cutometer MPA 580. For comparison of different locations on the body, back of the hand (left and right) and dorsal forearm (left and right) will be assessed for every participant at one time point (Visite 1).

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Distler, Prof.Dr.med, Principal Investigator — Department of Rheumatology
Locations (1):
- Department of Rheumatology, University Hospital Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Muller B, Ruby L, Jordan S, Rominger MB, Mazza E, Distler O. Validation of the suction device Nimble for the assessment of skin fibrosis in systemic sclerosis. Arthritis Res Ther. 2020 Jun 3;22(1):128. doi: 10.1186/s13075-020-02214-y. PMID 32493508